CLINICAL TRIAL: NCT01443065
Title: MEGA (Met or EGFR Inhibition in Gastroesophageal Adenocarcinoma): FOLFOX Alone or in Combination With AMG 102 or Panitumumab as First-line Treatment in Patients With Advanced Gastroesophageal Adenocarcinoma FNCLCC-FFCD-AGEO PRODIGE 17-ACCORD 20 Randomized Phase II Trial
Brief Title: MEGA (Met or EGFR Inhibition in Gastroesophageal Adenocarcinoma): FOLFOX Alone or in Combination With AMG 102 or Panitumumab as First-line Treatment in Patients With Advanced Gastroesophageal Adenocarcinoma
Acronym: MEGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRODIGE 17 / ACCORD 20/0904; 2009-012797-12 (EudraCT Number)
Record Dates: First submitted 2011-08-11; First posted 2011-09-29 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Malignant Neoplasm of Esophagus; Malignant Neoplasm of Stomach
Keywords: Adenocarcinoma; Locally advanced (non operable) or metastatic; First line treatment
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma | interventions — Oxaliplatin; Leucovorin; Panitumumab; rilotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A : simplified Folfox 4 (Active Comparator): Every 2 weeks :
  * Oxaliplatin : 85 mg/m2 over 120 mn (2h) IV on D1
  * Folinic acid : 400 mg/m² (racemic form) (or 200 mg/m² if L-folinic acid) over 2 h IV on D1 followed by :
  * 5-fluoro-uracil : 400 mg/m² in IV bolus on D1 followed by :
  * 5-fluoro-uracil : 2400 mg/m² in IV infusion over 46 h
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-fluoro-uracil
- Arm B : simplified FOLFOX 4 + panitumumab (Experimental): Every 2 weeks :
  * Oxaliplatin : 85 mg/m2 over 120 mn IV on D1
  * Folinic acid : 400 mg/m² (racemic form) (or 200 mg/m² with L-folinic acid) over 2 h IV on D1 (in Y to oxaliplatin) followed by :
  * 5-fluoro-uracil : 400 mg/m², IV bolus on D1, followed by :
  * 5-fluoro-uracil : 2400 mg/m², IV infusion IV over 46 h
  * Panitumumab : 6 mg/kg de 60 à 90 mn ± 15 mn IV every 14 days, just before chemotherapy administration (oxaliplatin and folinic acid), on Day 1 of each cycle. If the 1st infusion of panitumumab is well tolerated, the next infusions can be administered over 30 ± 10 mn.
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-fluoro-uracil; Drug: panitumumab
- Arm C : simplified FOLFOX 4 + AMG 102 (Experimental): Every 2 weeks :
  * Oxaliplatin : 85 mg/m2 over 120 mn IV on D1
  * Folinic Acid : 400 mg/m² (racemic) (or 200 mg/m² with L-folinic acid) over 2 h IV on D1 (in Y/concomitant with oxaliplatin) followed by :
  * 5-fluoro-uracil : 400 mg/m² IV bolus on D1 followed by :
  * 5-fluoro-uracil : 2400 mg/m² in IV perfusion over 46 h
  * AMG 102 : 10 mg/kg over 60 ± 15 mn IV every 14 days, just before chemotherapy administration (oxaliplatin and folinic acid), on Day 1 of each cycle. If the first infusion is well tolerated (without severe infusion-related reactions), the following infusions can be administered over 30 ± 10 mn.
  Interventions: Drug: Oxaliplatin; Drug: Folinic Acid; Drug: 5-fluoro-uracil; Drug: AMG102

INTERVENTIONS:
Drug: Oxaliplatin — 85mg/m² over 120 mn every 2 weeks up to progression or toxicity
  Other Names: Eloxatine
Drug: Folinic Acid — 400mg/m² over 120 mn every 2 weeks up to progression or toxicity
Drug: 5-fluoro-uracil — 400mg/m² in bolus, then 2400mg/m² over 46 h every 2 weeks up to progression or toxicity
Drug: panitumumab — 6mg/kg over 60-90 mn every 2 weeks up to progression or toxicity
  Other Names: Vectibix
  Arms: Arm B : simplified FOLFOX 4 + panitumumab
Drug: AMG102 — 10mg/kg over 60 mn every 2 weeks up to progression or toxicity
  Other Names: Rilotumumab
  Arms: Arm C : simplified FOLFOX 4 + AMG 102

SUMMARY:
This multicentre, open-label, randomized phase II trial is ongoing in 30 centres in France. Main eligibility criteria include: histologically proven adenocarcinoma of the stomach, esophagus or gastroesophageal junction; locally advanced or metastatic disease; measurable disease (RECIST 1.1); no known HER2 overexpression; no prior palliative chemotherapy.

DETAILED DESCRIPTION:
Patients are randomised to modified FOLFOX6 (oxaliplatin 85 mg/m2, FA 400 mg/m², FU 400 mg/m² bolus then 2400 mg/m² over 46 hr) alone or combined to either panitumumab (6 mg/kg) or AMG 102 (10 mg/kg), every two weeks until unacceptable toxicity or disease progression. Judgment criteria include 4-month progression-free survival (PFS) rate (primary endpoint), OS, objective response rate, and safety. Ancillary studies aim to identify candidate predictive and prognostic biomarkers among functional of molecular alterations of the EGFR/RAS/RAF and HGF/c-Met pathways, and to monitor circulating tumour cells and circulating immune cells (myeloid derived suppressor cells, NK cells) in sequential blood samples taken at baseline and through the study treatment. A total of 165 pts will be enrolled (Fleming's one-step design)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach, the esophagus or the cardia (with or without signet ring cells; intestinal, diffuse or mixed form).
* Locally advanced (non resectable) or metastatic disease.
* Measurable disease (at least one measurable tumor) according to the RECIST V1.1 criteria (the tumor should not be located in a previous field of radiation).
* Absence of previous palliative chemotherapy. Previous neo-adjuvant or adjuvant chemotherapies (alone or combinated with radiotherapy) are authorized, including biotherapy (except anti-EGFR or anti-c-Met / HGF), if it has been stopped at least 12 months before inclusion.
* Previous radiotherapy authorized if stopped at least 14 days before randomization and if at least one measurable target outside the radiation area is present.
* No major surgery ≤ 28 days, or minor surgery ≤ 14 days, prior to randomization
* Sites of disease evaluated within 28 days prior to randomization with thoracic-abdominal-pelvic CT scan (or abdominal-pelvic MRI plus Chest X-ray).
* Age ≥ 18 years.
* Patient general status : ECOG 0-1.
* Life expectancy ≥ 3 months.
* Hemoglobin > or = 9 g/L - (transfusion authorized if necessary), PNN ≥ 1,5.109/l, platelets ≥ 100.109/l.
* Hepatic transaminases ≤ 2.5 times upper limit of normal (ULN) (≤ 5 ULN in case of hepatic metastases), alkaline phosphatase ≤ 2.5 ULN (≤ 5 ULN in case of hepatic metastases), total bilirubinemia ≤ 1.5 ULN)
* Creatinine clearance (calculated or measured) ≥ 50 ml / min, serum creatinine > 1.5 ULN
* Prothrombin time (PT) ≥ 60 %, INR < 1,5 (except if anticoagulant therapy)
* Magnesemia and calcemia ≥ Lower Limit of Normal (LLN)
* Negative Pregnancy test for women of child-bearing age.
* Information given to the patient and signed informed consent.
* Public Health insurance coverage.
* Sample of tumour (primitive or metastatic) available.

Exclusion Criteria:

* Known brain or leptomeningeal metastases.
* Positive HER2 Status (IHC 3+ or IHC2+/FISH or CISH+) .
* contraindication, allergy or hypersensitivity to ANY OF the study treatments.
* Prior Treatment with EGFR inhibitor or HGF / c-Met inhibitor.
* Patient already included in another clinical trial testing an experimental drug.
* Peripheral edema > grade 2.
* Proteinuria > 1 g/24h
* Clinically significant cardiovascular disease (such as unstable angina pectoris, severe congestive heart failure, uncontrolled severe cardiac arrhythmia) within 12 months prior to randomization.
* Thrombosis or ischemic vascular event during the last 12 months (deep venous thrombosis, pulmonary embolism, STROKE or established cerebral infarction, myocardial infarction).
* Medical history or signs of interstitial pneumopathy or pulmonary fibrosis.
* Peripheral neuropathy > grade 1.
* Clinically significant hemorrhage of the upper gastrointestinal tract (requiring blood transfusion or hemostatic interventional procedure.
* Actively evolutive inflammatory bowel disease or any other intestinal disease causing chronic diarrhea (≥ grade 2).
* Any uncontrolled concomitant disease (e.g., uncontrolled diabetes) or medical history (e.g., organ transplantation) which, according to the opinion of the investigator, may interfere with the interpretation of the study results.
* Any comorbidity or situation which, according to the opinion of the investigator, could increase the risk of toxicity (e.g., Dihydropyrimidine dehydrogenase deficiency).
* Chronic or active HIV, HBV or HCV infections.
* Severe and\or not healed wound.
* Any active infection requiring systemic treatment, or any uncontrolled infection within 14 days before randomization.
* Other concomitant malignancy or history of cancer (except carcinoma in situ of the cervix, or non melanoma skin cancer, with curative intent treatment), except when considered in complete remission for at least 5 years before randomization.
* Pregnant women or women who might become pregnant during the study (or who plan to become pregnant within 6 months after the last administration of a study drug) or lactating women.
* Men or women who have the age of procreation and who do not abide with the use of a highly efficient contraceptive means (according to the current institutional standards) or, alternatively, the use of abstinence during the study treatment and until 6 months after last administration of the study drugs.
* Patient unwilling to comply with the medical follow-up required by the trial because of geographic social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 4 months | 4 months
  based on the proportion of success in each patient group (patient without progression at 4 months)

SECONDARY OUTCOMES:
Progression-free survival | until progression or death
  Progression-free survival is defined as the time from randomization to progression (RECIST v1.1 criteria) or death. Patients alive without progression will be censored at the last tumoral evaluation and 5 years maximum.
Overall survival | until death
  Overall survival is defined as the time from randomization to death any cause or last follow-up news (censored data).
Time to progression | 4 months
  Time to progression is defined as the time from randomization to progression (RECIST v1.1 criteria). Patients alive without progression will be censored at the last tumoral evaluation. Patients died without progression will be censored at the death date any cause.
Objective tumor response rate (OR) (= complete responses [CR] + partial responses [PR]) according to RECIST V1.1 | until progression
  The objective tumor response will be evaluated by the investigator with RECIST v1.1 criteria every 8 (± 1) weeks up to disease progression. Patients with symptoms suggestive of disease progression will have a tumoral evaluation when symptoms will occur.
Objective response duration | until progression
  The Objective response duration is defined as time from first Complete Response or Partial Response to progression. Patients died without progression will be censored at death date.
Disease control rate (Complete Response + Partial Response + stable disease [SD]) | 4 months
  The tumor control rate is rate of objective responses (complete responses and partial responses) and stable disease responses.
Tolerance of the treatment | 24 months
  Tolerability of the treatment will be based on toxicities of evaluated products by clinical and biological measurements (NCIC/CTC (CTCAE V4) criteria, except for peripheral neuropathy toxicity (Lévi scale)).

CONTACTS AND LOCATIONS:
Overall Officials: David MALKA, Dr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Eric FRANCOIS, Dr, Principal Investigator — Centre Antoine Lacassagne, Nice; Bruno BUECHER, Dr, Principal Investigator — Institut Curie Paris; Christophe BORG, Pr, Principal Investigator — Hôpital Andre Boulloche-MONTBELIARD; Emmanuelle SAMALIN, Dr, Principal Investigator — Centre Val d'Aurelle Paul Lamarque-MONTPELLIER; You Heng LAM, Dr, Principal Investigator — Centre Paul Papin-ANGERS; François GHIRINGHELLI, Dr, Principal Investigator — Centre Georges Francois Leclerc-DIJON; Driffa MOUSSATA, Dr, Principal Investigator — Centre Hospitalier Lyon Sud-PIERRE BENITE; Marie-Pierre GALAIS, Dr, Principal Investigator — Centre Francois Baclesse-CAEN; Frédérique CVITKOVIC, Dr, Principal Investigator — Centre René Huguenin-SAINT-CLOUD; Marie-Claire KAMINSKY, Dr, Principal Investigator — Centre Alexis Vautrin-VANDOEUVRE LES NANCY; Olivier BOUCHE, Pr, Principal Investigator — Hôpital Robert Debré - REIMS; Julien TAIEB, Pr, Principal Investigator — Hôpital Européen Georges Pompidou-PARIS (HEGP); Cédric LECAILLE, Dr, Principal Investigator — Polyclinique Bordeaux Nord Aquitaine-BORDEAUX; Yves BECOUARN, Dr, Principal Investigator — Institut Bergonié Bordeaux; Barbara DAUVOIS, Dr, Principal Investigator — Centre Hospitalier La Source-ORLEANS; Julien FORESTIER, Dr, Principal Investigator — Hôpital Edouard Herriot-LYON; Jaafar BENNOUNA, Dr, Principal Investigator — Centre René Gauducheau; Christelle DE LA FOUCHARDIERE, Dr, Principal Investigator — Centre Leon Berard; Christophe BORG, Pr, Principal Investigator — Centre Hospitalier Jean Minjoz; Jean Baptiste BACHET, Dr, Principal Investigator — Centre Hospitalier La Pitié Salpétrière; Jean Luc RAOUL, Dr, Principal Investigator — Institut Paoli-Calmettes; Leila BENGRINE LEFEVRE, Dr, Principal Investigator — Hôpital Saint Antoine; Laurent MIGLIANICO, Dr, Principal Investigator — CHP Saint Grégoire; Laetitia DAHAN, Dr, Principal Investigator — Centre Hospitalier La Timone; Thomas APARICIO, Pr, Principal Investigator — Hôpital Avicenne; Hervé PERRIER, Dr, Principal Investigator — Hôpital Saint Joseph; Jean Philippe METGES, Dr, Principal Investigator — CHU Morvan; Eric TERREBONNE, Dr, Principal Investigator — Hôpîtal haut Lévèque; Pascal ARTRU, Dr, Principal Investigator — Hôpital Privé Jean Mermoz; Gaël DEPLANQUE, Dr, Principal Investigator — Groupe Hospitalier Saint Joseph; Emmanuel MAILLARD, Dr, Principal Investigator — CHR Annecy; Antoine ADENIS, Pr, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Institut Gustave Roussy, Villejuif, France